CLINICAL TRIAL: NCT00550212
Title: An Open-Label, Single-Dose Study of the Mass Balance and Metabolic Disposition of Orally Administered [14C]-Labeled HKI-272 in Healthy Male Subjects
Brief Title: Study Evaluating Oral Administrations of HKI-272 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3144A1-1108
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: healthy subjects
MeSH Terms: interventions — neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 240 mg
  Interventions: Drug: neratinib

INTERVENTIONS:
Drug: neratinib — HKI-272, Single-dose capsule and solution

SUMMARY:
The purpose of this study is to evaluate the mass balance and metabolic distribution of C14-labeled HKI-272 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, aged 18 to 50 years.

Exclusion Criteria:

* Female subjects

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Mass balance, metabolic distribution, PK | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology